CLINICAL TRIAL: NCT03203447
Title: A Randomized, Masked, Controlled Trial To Study The Safety And Efficacy Of Suprachoroidal CLS-TA In Combination With An Intravitreal Anti-VEGF Agent In Subjects With Retinal Vein Occlusion
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide With IVT Anti-VEGF in Subjects With Macular Edema Following RVO
Acronym: TOPAZ
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The early termination is due to the results obtained from the sister study, SAPPHIRE (CLS1003-301), which did not meet the 8-week primary efficacy endpoint.
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLS1003-302
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: RVO; ME; Microneedle; Microinjection; Triamcinolone; Choroid; Choroid injection; Suprachoroidal; Anti-VEGF; Subretinal Fluid; Cystoid Macular Edema; Optical Coherence Tomography; OCT; Central Subfield Thickness; Lucentis; Avastin; Ranibizumab; Bevacizumab; Triamcinolone acetonide
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Triamcinolone Acetonide; Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Lucentis (0.5 mg/0.05 mL), IVT injection + CLS-TA (4 mg/0.10 mL), SC injection or Avastin (1.25 mg/0.05 mL), IVT injection + CLS-TA (4 mg/0.10 mL), SC injection
  Interventions: Drug: suprachoroidal CLS-TA; Drug: Lucentis or Avastin
- Control (Sham Comparator): Lucentis (0.5 mg/0.05 mL), IVT injection + sham SC procedure or Avastin (1.25 mg/0.05 mL), IVT injection + sham SC procedure
  Interventions: Drug: suprachoroidal sham; Drug: Lucentis or Avastin

INTERVENTIONS:
Drug: suprachoroidal CLS-TA — suprachoroidal injection of CLS-TA
  Other Names: Triamcinolone acetonide
  Arms: Active
Drug: suprachoroidal sham — sham suprachoroidal procedure
  Arms: Control
Drug: Lucentis or Avastin — IVT anti-VEGF agent. Either a 0.5 mg intravitreal injection of Lucentis or 1.25 mg intravitreal injection of Avastin
  Other Names: IVT anti-VEGF agent

SUMMARY:
This Phase 3, multicenter, randomized, masked, controlled, parallel group study is designed to demonstrate that suprachoroidal (SC) CLS-TA administered with intravitreal (IVT) anti-VEGF agent in subjects with treatment naive RVO is superior to IVT anti-VEGF agent used alone.

DETAILED DESCRIPTION:
A Randomized, Masked, Controlled Trial to Study the Safety and Efficacy of Suprachoroidal CLS-TA With Intravitreal Anti-VEGF Agent in Subjects With Retinal Vein Occlusion

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of RVO in the study eye
* Has a CST of ≥ 300 µm in the study eye
* Has an ETDRS BCVA score of ≥ 20 letters read and ≤ 70 letters read in the study eye
* Is naïve to local pharmacologic treatment for RVO in the study eye

Exclusion Criteria:

* Any active ocular disease or infection in the study eye other than RVO
* History of glaucoma, intraocular pressure > 21 mmHg or ocular hypertension requiring more than one medication
* Any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study
* Any evidence of neovascularization in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Chief Medical Officer
Locations (92):
- United States (72):
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Centers PC, Tucson, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Win Retina, Arcadia, California
  - Retina Vitreous Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Retina Consultants of Orange County, Fullerton, California
  - Macula and Retina Institute, Glendale, California
  - American Institute of Research, Los Angeles, California
  - Retina Vitreous Associates Medical Group Inc, Mountain View, California
  - Stanford University - Byers Eye Institute, Palo Alto, California
  - Retina Consultants of Southern California, Redlands, California
  - Retina Consultants Medical Group Inc, Sacramento, California
  - American Institute of Research, Whittier, California
  - Retina Group of New England, PC, New London, Connecticut
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Specialty Retina Center, Coral Springs, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Center for Retina Care at The Eye Institute, Melbourne, Florida
  - Florida Retina Institute, Orlando, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - East Florida Eye Institute EFEI, Stuart, Florida
  - Southern Vitreoretinal Association, Tallahassee, Florida
  - Center for Retina And Macular Disease, Winter Haven, Florida
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Gailey Eye Clinic, Bloomington, Illinois
  - University and Macula Associates, Oak Forest, Illinois
  - Prairie Eye Center, Ltd., Springfield, Illinois
  - Sabates Eye Centers, Leawood, Kansas
  - Vitreo-Retinal Consultants and Surgeons PA, Wichita, Kansas
  - Central Plains Eye MDs, Wichita, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Retina Specialists, Baltimore, Maryland
  - The Retina Care Center, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - The National Retina Institute, Towson, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Associated Retinal Consultants PC, Grand Rapids, Michigan
  - Vitreo-Retinal Associates, P.C., Grand Rapids, Michigan
  - Associated Retinal Consultants P.C., Royal Oak, Michigan
  - Retina Consultants of Michigan, Southfield, Michigan
  - Associated Retinal Consultants PC, Traverse City, Michigan
  - Retina Associates of St. Louis, Florissant, Missouri
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Retina Associates of Western New York, Rochester, New York
  - Island Retina, Shirley, New York
  - Retina-Vitreous Surgeons of Central New York, Syracuse, New York
  - Retina Associates of Cleveland Inc, Middleburg Heights, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Pennsylvania Retina Specialists PC, Camp Hill, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Texas Retina Associates - Arlington, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina and Vitreous of Texas, PLLC, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Retina Specialists, Plano, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of South Texas PA, San Antonio, Texas
  - Retina Consultants of Houston, PA, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Retina Group of Washington, Fairfax, Virginia
  - West Virginia University Medicine Eye Institute, Morgantown, West Virginia
- Australia (3):
  - Eye Clinic Albury Wodonga, Albury, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Save Sight Institute, University of Sydney (Sydney Eye Hospital), Sydney, New South Wales
- MH EK Honvédkórház, Budapest, Hungary
- India (15):
  - Raghudeep Eye Hospital, Gujrāt, Ahmedabad
  - LV Prasad Eye Institute, Hyderabad, Andhra Pradesh
  - L V Prasad Eye Institute, Visakhapatnam, Andhra Pradesh
  - R.P. Centre, AIIMS, New Delhi, Ansari Nagar
  - Narayana Nethralaya, RajajiNagar, Bangalaore
  - LV Prasad Eye Institute, Pātia, Bhubaneswar
  - M&J Western Regional Institute of Ophthalmology, Asarwa, Gujarat
  - PBMA's H.V Desai Eye Hospital, Pune, Maharashtra
  - Dr Shroff 's Charity Eye Hospital, Delhi, New Delhi
  - Regional Institute of Ophthalmology, Bihār, Patna
  - B B Eye Foundation VIP, Kolkata, Raghunathpur
  - SMS Hospital, Jaipur, Rajasthan
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Jawaharlal Rohatgi Eye Hospital, Kanpur, Uttar Pradesh
  - Disha Eye Hospitals Pvt. Ltd., Kolkata, West Bengal
- Auckland Eye, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 162 (Two patients were randomized to the Active arm, but did not receive study drug.) | 163 (One patient was randomized to the Control arm, but did not receive study drug.)
Completed | 0 | 0
Not Completed | 162 | 163
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 10
Not completed — Includes premature discontinuation due to study termination and unknown | 159 | 152

BASELINE CHARACTERISTICS:
Population: The Safety population included all randomly assigned subjects who were administered at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 160 | 162 | 322
Age, Categorical [Count of Participants; unit: Participants] — Age of patients in years relative to the date of the Screening visit.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 75 | 91 | 166
    >=65 years | 85 | 71 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of patients in years relative to the date of the Screening visit.
  years | 63.8 (13.07) | 62.6 (12.26) | 63.2 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 93 | 172
  Male | 81 | 69 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 72 | 70 | 142
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 6 | 3 | 9
  White | 77 | 84 | 161
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 2 | 0 | 2
  United States | 96 | 98 | 194
  Australia | 2 | 3 | 5
  India | 60 | 61 | 121
Type of Retinal Vein Occlusion [Count of Participants; unit: Participants]
  Branch retinal vein occlusion | 90 | 93 | 183
  Central retinal vein occlusion | 70 | 69 | 139

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Demonstrating ≥ 15 Letter Improvement From Baseline in Early Treatment of Diabetic Retinopathy Study (ETDRS)
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on an ETDRS eye chart. An increase from the pre-treatment state in BCVA of 15 letters or more represents a clinically meaningful improvement.
Time Frame: 2 months
Population: The Intent-to-treat population included all randomized patients. Values for missing data were imputed using last observation carried forward.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 162 | 163
Participants | 64 | 76
Statistical Analysis 1: Comparison: Active vs Control; Based on a Pearson chi-square test, a total sample size of approximately 460 subjects provided 90% power to detect a difference of 15% between the Active and Control arms assuming the Control arm showed a proportion of 0.50 at 8 weeks. The primary analysis was a test of superiority of the Active arm over the Control arm, and was based on a Cochran-Mantel-Haenszel chi-square test stratified by type of retinal vein occlusion; Test type: Superiority; p = 0.191, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance was 0.050. Prior to evaluating the results of the CMH test, a Breslow-Day test with Tarone's adjustment was conducted to confirm the homogeneity of the odds ratios between RVO strata; The CMH test was stratified by the type of retinal vein occlusion, i.e., branch vs. central; Difference in percentages = -7.1, 95% CI 2-sided [-17.9 to 3.6] — Estimated value was calculated as the percentage of subjects in the Active arm meeting the primary endpoint minus the percentage of subjects in the Control arm meeting the primary endpoint

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on an ETDRS eye chart. A positive change from baseline value represents an improvement in vision.
Time Frame: 6 months
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment. Values for missing data were not imputed.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 160 | 159
letters | 13.8 (1.96) | 20.7 (1.91)

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A masked reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema.
Time Frame: 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | Active | Control
Number analyzed (Participants) | 162 | 159
microns | -353.6 (19.60) | -374.7 (19.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through follow-up and study completion, approximately 6 months.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/162
Serious Adverse Events (participants affected / at risk) | 1/160 | 3/162
Other Adverse Events (participants affected / at risk) | 11/160 | 1/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=160) | Control (N=162)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=160) | Control (N=162)
Intraocular pressure increased (Investigations) | 11 (14) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early termination of the trial by sponsor, 325 of the planned 460 were enrolled. All planned study visits were not completed by all treated subjects; therefore, all planned data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03203447/Prot_SAP_000.pdf